CLINICAL TRIAL: NCT07067827
Title: Clinical Validation of a Self-questionnaire in Adults With Osteoporosis
Brief Title: Self-questionnaire in Osteoporosis
Status: Recruiting | Type: Observational
Sponsor: CHU de Quebec-Universite Laval (Other)
Responsible Party: Sponsor
Other Study IDs: 2026-8073
Record Dates: First submitted 2025-07-07; First posted 2025-07-16 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Osteoporosis
Keywords: osteoporosis; self-administered questionnaire; family history; rare genetic bone diseases
MeSH Terms: conditions — Osteoporosis | interventions — Pedigree

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group starting with the self-administered questionnaire followed by the family tree and vice versa: Recruited patients will be randomized to either start with the self-administered questionnaire or the family tree. Then, 3 months later, those who started with the questionnaire will be able to do the interview for the family tree and vice versa.
  Interventions: Other: Self-administered questionnaire; Other: Family tree

INTERVENTIONS:
Other: Self-administered questionnaire — The self-administered questionnaire was previously prepared by the research team for another project. It includes 14 questions addressing the dentition, fractures, joint hypermobility, height, and eye abnormalities present in the participants or their relatives. This questionnaire covers the clinical manifestations of rare bone diseases such as osteogenesis imperfecta, pycnodysostosis, hypophosphatasia, and osteopetrosis. This self-administered questionnaire will be filled online by participant. Average completion time of 20 minutes.
Other: Family tree — For the family tree, this step is done by a telephone interview lasting a maximum of 45 minutes, depending on the size of the participant's family. The researcher will be able to reconstruct the family history with the index case. The family tree will then contain the family history up to the second degree of kinship with respect to the index cases. The information collected through the index cases when creating the family tree must include, for each relative, biological sex, as well as information on the presence or absence of a rare or genetic bone disease and clinical signs associated with these diseases, such as short stature, bone deformities, deafness, eye problems, etc.

SUMMARY:
Osteoporosis is a multifactorial disease in which genetic predispositions play a key role in its development. A better understanding of family history and clinical manifestations among first- and second-degree relatives can help improve early detection and personalized care for at-risk patients. To this end, we will test a self-administered questionnaire previously developed by our research team. This questionnaire includes the main manifestations associated with rare genetic bone diseases such as osteogenesis imperfecta, hypophosphatasia, and osteopetrosis.

DETAILED DESCRIPTION:
The main objective of this project is to test the validity of this new self-administered questionnaire, by studying the concordance between its answers and those obtained from a patient's family tree by telephone.

Primary Objective: To test the validity of a self-administered questionnaire to facilitate the identification of rare genetic bone diseases in adults with osteoporosis.

Secondary Objectives: To adapt the self-administered questionnaire to increase the accuracy of responses compared to those obtained using a family tree, with the aim of using it for clinical screening of rare genetic bone diseases in adults.

Data collection:

Sociodemographic data (age, sex, ethnicity, body mass index, menopausal status, smoking, alcohol consumption, physical activity, history of falls in the past year) and clinical data will be collected from participants' electronic medical records at the CHU de Québec-Université Laval (age at osteoporosis diagnosis, history of osteoporotic fractures, osteoporosis risk category based on the most recent bone density scan, calcium and/or vitamin D supplement use, history of anti-osteoporosis medications, presence of comorbidities, use of prednisone or antihormonal medications) to describe the participants and the severity of their osteoporosis. Other data collection will be conducted in two stages. First, recruited patients will be randomized to either begin with the self-administered questionnaire or the family tree. Then, 3 months later, the people who started with the questionnaire will be able to do the interview for the family tree and vice versa.

Randomization: For this collection, a balanced block randomization will be used to randomly assign patients to one of the two assessment administration sequences. This approach, which corresponds to a crossover design with sequence randomization, will balance order effects and ensure a similar distribution in each sequence. In addition, the use of blocks (of size 4) will ensure that the balance between the two conditions is maintained throughout the recruitment period.

Statistical analyzes:

Descriptive statistics will first be performed to characterize the participants (age, sex, number of first- and second-degree relatives, as well as the clinical manifestations detailed in the self-administered questionnaire) and to report, based on the relationship, the frequency of different clinical manifestations in relatives. In this study, the pedigree will serve as the gold standard to describe the presence or absence of familial bone disease, specifying the degree of affected kinship, the type of inheritance, and the most likely diagnosis (e.g., hypophosphatesia, osteogenesis imperfecta, etc.). The concordance between the responses provided by the self-administered questionnaire and the information from the pedigree will be primarily assessed by calculating the kappa coefficient. This analysis will constitute the primary statistical approach of the study. In addition, secondary analyses will be conducted to determine the sensitivity and specificity of the self-administered questionnaire compared to the gold standard. These measurements will make it possible to evaluate the diagnostic performance of the tool developed in the detection of familial bone disease.

Sample size calculation: The agreement between the two assessment tools will be based mainly on questions with three response categories (Yes, No, Don't know) with respective frequencies assumed to be (0.1, 0.3 and 0.6). The objective being to test whether the agreement, measured by the kappa coefficient, exceeds the threshold of 0.7 (H0: Kappa ≤ 0.7 versus H1: Kappa > 0.7), the comparison will be carried out using a one-sided Z-test for kappa, setting the type I error rate (α) at 0.05. To detect a kappa coefficient of 0.9 with a power of 80%, it is necessary to recruit 58 patients. The sample size was calculated using PASS 2024 software, version 24.0.2.

ELIGIBILITY:
Inclusion Criteria:

* Adult over 18
* Followed by the rheumatology or endocrinology clinics at the CHUL (CHU de Quebec-Universite Laval)
* Suffer from osteoporosis
* Have internet access

Exclusion Criteria:

* Unfit, unable to consent, unable to answer a questionnaire, unknown family history (e.g. adopted person)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults followed at the rheumatology and endocrinology clinic of the CHUL in Quebec
Sampling Method: Probability Sample
Enrollment: 58 (Estimated)
Dates: Start 2025-07-30 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Concordance between the results of the self-questionnaire compared to those obtained by a family tree. | 3 months
  Descriptive statistics will first be performed to characterize the participants (age, sex, number of first- and second-degree relatives, as well as the clinical manifestations detailed in the self-administered questionnaire) and to report, based on the relationship, the frequency of different clinical manifestations in relatives. In this study, the pedigree will serve as the gold standard for describing the presence or absence of familial bone disease, specifying the degree of affected kinship, the type of inheritance, and the most likely diagnosis (e.g., hypophosphatasia, osteogenesis imperfecta, etc.).
  The concordance between the responses provided by the self-administered questionnaire and the information from the pedigree will be primarily assessed by calculating the kappa coefficient. This analysis will constitute the main statistical approach of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Laetitia Michou, MD PhD, Principal Investigator — CHU de Quebec-Universite Laval
Locations (1):
- CHU de Quebec-Universite Laval, Québec, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided